CLINICAL TRIAL: NCT05039346
Title: Quality of Life and Patient Needs in Advanced High Grade Gliomas - A Prospective Study
Brief Title: Quality of Life and Patient Needs in Advanced High Grade Gliomas
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Tobias Walbert, MD, PhD, Co-Director Hermelin Brain Tumor Center at the Henry Ford Cancer Institute, Henry Ford Health System
Other Study IDs: IRB 14537
Record Dates: First submitted 2021-08-27; First posted 2021-09-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Quality of Life; Brain Tumor; Glioblastoma; Glioma; Anaplastic Astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Glioma; Astrocytoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain Tumor: Patients who are diagnosed with a high grade glioma that is progressive and therapy resistance. Patients will have a KPS of 60 or less.
  Interventions: Other: Phone interviews
- Care Giver: Should a patient be unable to answer, the care giver will step in and provide surrogate answers.
  Additionally, at four weeks following the patient's death, the patient's care giver will be interviewed by utilizing a validated questionnaire.
  Interventions: Other: Phone interviews

INTERVENTIONS:
Other: Phone interviews — Phone interviews will be used to determine the patient's quality of life, symptoms and performance status

SUMMARY:
There is limited knowledge regarding the quality of life and needs of patients with advanced high grade gliomas, especially during the end of life. By doing this research, we are able to assess caregiver and patient symptoms and needs during the end of life phase of patients with brain tumors.

DETAILED DESCRIPTION:
Purpose: This is a pilot study to prospectively assess the symptoms and quality of life of patients and with advanced high grade glioma and their care takers.

Specific Aims: The aim of this study is to investigate the symptoms of patients with advanced high grade glioma. Patients who failed 3rd line chemotherapy and who require at least occasional assistance will be prospectively followed and their symptoms will be prospectively assessed. Patient's caregiver will be interviewed following the death of the patient to assess clinical symptoms in the last weeks of life and around the time of death.

Methods: Patients will undergo clinical symptom assessment via questionnaire. Patients will be followed by regular semi-structured phone interviews.

Should a patient pass, four weeks following this, the patient's care giver will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Tissue proven diagnosis of a high grade brain tumor
* Disease progression by MRI
* Therapy resistant tumor to 2nd line chemotherapy
* Karnofsky Performance Scale (KPS) score of 60 or less
* Patient will need to assign caregiver

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been diagnosed with a high grade brain tumor and must show signs of clinical progression. Patients who have failed 3rd line chemotherapy regimen and who require at least occasional assistance are invited to participate.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-02-11 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Quality of life and end of life symptoms in brain tumor patients | 12 months
  Assessment will be performed with validated questionnaire (MDASI-BT)
Examination | 12 months
  Clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Walbert, MD, PhD, Principal Investigator — Henry Ford Health System

IPD SHARING:
Plan to Share IPD: No